CLINICAL TRIAL: NCT05284669
Title: Effect of an E-learning Intervention on Knowledge, Attitudes and Beliefs of Healthcare Professionals Managing Low Back Pain: a Randomized Controlled Trial With Nested Process Evaluation.
Brief Title: Effect of an E-learning Intervention on Knowledge, Attitudes and Beliefs of Healthcare Professionals Managing Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antoine Fourré (Other)
Collaborators: University of Mons (Other); Universiteit Antwerpen (Other); Universite de Picardie Jules Verne (Other)
Responsible Party: Sponsor-Investigator, Antoine Fourré, PhD student - Research Assistant, Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20/51/714
Record Dates: First submitted 2022-03-10; First posted 2022-03-17 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Knowledge, Attitudes, Practice; Low Back Pain; Physical Therapy; Physicians
Keywords: Distance education; Musculoskeletal pain; Guideline adherence; First-line care
MeSH Terms: conditions — Behavior; Low Back Pain; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental e-learning (Experimental): The experimental interactive intervention is based on international guidelines for the management of LBP and includes multiple interactions with the participant in a virtual environment. Metaphors and concrete clinical situations are presented to translate the knowledge (i.e. the management of low back pain from a biopsychosocial point of view) to clinical practice. Interactions consists of videos, open and closed questions and audio records.
  Interventions: Other: Experimental e-learning
- Traditional e-learning (Other): The traditional intervention consists of a traditional online lecture based on international guidelines for the management of LBP without any interaction. The focus is more fundamental (theoretical) without metaphors or clinical cases.
  Interventions: Other: Traditional e-learning

INTERVENTIONS:
Other: Experimental e-learning — Interactive lecture based on the guidelines for the management of LBP with a focus on self-management and patient's reassurance
  Arms: Experimental e-learning
Other: Traditional e-learning — Traditional lecture based on the guidelines for the management of LBP with a focus on diagnostic triage and specific cause of LBP
  Arms: Traditional e-learning

SUMMARY:
The purpose of the current research project is to examine if the healthcare professionals (HCPs) knowledge, attitudes, beliefs and behavior about the management of low back pain (LBP) patients changes following an e-learning intervention (experimental interactive e-learning versus traditional non-interactive e-learning)

DETAILED DESCRIPTION:
The purpose of the current research project is to use an e-learning educational approach to implement guideline-adherent care in first line HCPs. We aim to enhance the knowledge, attitudes, beliefs and behavior of HCPs towards a biopsychosocial approach in the management of LBP patients. We will compare the effect of an interactive e-learning intervention (i.e. experimental intervention) to an e-learning intervention without interaction (i.e. traditional intervention). Both interventions will be based on the most recent scientific literature regarding the management of LBP, but both the focus and the didactical approach will slightly differ between the interventions. We will use a mixed methods approach to gain an in-depth understanding of HCPs behavior in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* To be an healthcare practitioner (general practitioner, physiotherapist, specialist physician, student in medicine including specialization, student in physiotherapy)
* Working or studying in Belgium or France
* Being in possession of an internet connected device (e.g. computer, tablet or smartphone) with speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2720 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
The Health Care Providers Pain and Impairment Relationship Scale (HC-PAIRS) | Baseline assessment and post-intervention assessment (between 2 and 4 weeks after baseline)
  The HC-PAIRS assesses attitudes and beliefs about functional expectations for patients with chronic LBP. It consists of 13 statements that must be rated on a seven-point Likert scale, ranging from 'totally disagree' to 'totally agree'. A high score on the HC-PAIRS reflects a belief with a strong relationship between pain and impairment. Psychometric properties of this questionnaire have been established.
Vignette of Rainville | Baseline assessment and post-intervention assessment (between 2 and 4 weeks after baseline)
  The clinical vignette described a patient with non-specific LBP. This vignette was developed by Rainville. Participants were asked to assess the patient's ability to work, from 1 (full-time) to 5 (remain out of work) and gave their opinion on the appropriate level of activity, with choices graded from 1 (no limitations on activity) to 5 (limit all physical activity). If the score of the participant was between 1 and 2 it was considered guideline adherent. If the score was between 3 and 5 it was considered guidelines discordant.

SECONDARY OUTCOMES:
The Back Pain and Attitudes Questionnaire (Back-PAQ ; 10-items version) | Baseline assessment and post-intervention assessment (between 2 and 4 weeks after baseline)
  The Back-PAQ questionnaire (10 items version) assesses attitudes and underlying beliefs about back pain on a 5-point Likert scale. The scoring of the answers ranges from -2 to +2. A negative score reflects beliefs that are unhelpful and vice-versa. All items were written in the second person to personalize the questionnaire. The purpose of this personalization is that HCPs or students present their own beliefs rather than projecting their beliefs onto people with LBP or presenting their beliefs about people with LBP.
The Neurophysiology of Pain Questionnaire (NPQ) | Baseline assessment and post-intervention assessment (between 2 and 4 weeks after baseline)
  The Neurophysiology of pain questionnaire (NPQ) assesses how an individual conceptualizes biological mechanisms underpinning pain. The NPQ includes 19 questions with three answer options (true; undecided; false). The scoring is 1 for a correct answer and 0 if the participant was wrong or undecided. This questionnaire was included to reflect recommendations of the guidelines for the management of LBP that encourages clinicians to explain and reassure the patient about their personal experience of pain.
Fictive clinical cases of patients with LBP | Baseline assessment and post-intervention assessment (between 2 and 4 weeks after baseline)
  4 clinical cases were developed by a multidisciplinary team of experts in the field (general practitioners, orthopedic surgeons, physiotherapists, and academics). Two cases described the symptoms of a patient with specific LBP and the two others described the symptoms of a patient with non-specific LBP. A specific and non-specific clinical case were presented at baseline and post-intervention assessment. Participants answered 3 open questions related to the clinical case: "In your opinion, what are the causes/contributing factors to the pain of this patient?"; "As an healthcare practitioners what would be your first approach to manage this patient?"; "Which advices would you give to this patient concerning physical activity".
  Coding of the answers in a matrix using keywords and themes will be used to analyse the orientation of the healthcare practitioners (guideline adherent or guideline discordant).
Experiences of HCPs with the e-learning (quantitative) | Post-intervention assessment (between 2 and 4 weeks after baseline)
  A Likert scale (1-7) will be used to examine the participants experiences regarding the content and quality of the intervention and the Technology acceptance. The questions of this survey are based on Cheng et al. 2012 and cover global system quality and technology acceptance of the e-learning. Higher score reflects a better experience with the e-learning intervention.
Experiences of HCPs with the e-learning (qualitative) | Between 4 and 6 weeks after baseline
  A purposive sample of participants agreeing to take part in a phone interview will be invited to an in-depth interview. We foresee to start with 10 HCPs of each group (experimental and traditional e-learning intervention) to provide depth and breadth of experiences and will continue until no new themes emerge (Bowen 2008). The principles of qualitative research will be used to explore how participants experienced the e-learning intervention and which impact had the e-learning on their clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Roussel, PhD, Principal Investigator — Universiteit Antwerpen; Laurence Ris, PhD, Study Director — University of Mons; Antoine Fourré, MSc, Principal Investigator — University of Mons / University of Antwerp; Rob Vanderstraeten, MSc, Principal Investigator — Universiteit Antwerpen; Jef Michielsen, MD, PhD, Study Director — Universiteit Antwerpen; Hilde Bastiaens, MD, PhD, Study Director — Universiteit Antwerpen; Sybil Anthierens, PhD, Study Director — Universiteit Antwerpen; Frédéric Telliez, PhD, Study Director — Universite de Picardie Jules Verne
Locations (1):
- Online study, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fourre A, Fierens A, Michielsen J, Ris L, Dierick F, Roussel N. An interactive e-learning module to promote bio-psycho-social management of low back pain in healthcare professionals: a pilot study. J Man Manip Ther. 2022 Apr;30(2):105-115. doi: 10.1080/10669817.2021.1988397. Epub 2021 Oct 22. PMID 34678129
- See also: Website of the European project (Interreg FWVl NOMADe - N° 4.7.360) — http://nomadeproject.eu